CLINICAL TRIAL: NCT04307472
Title: Leveraging the Electronic Health Record to Nudge Clinicians to Prescribe Evidence-Based Statin Medications to Reduce the Risk of Cardiovascular Disease: A Randomized Clinical Trial
Brief Title: Nudges for Statin Prescribing in Primary Care
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Collaborators: National Institute on Aging (NIA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Double | Purpose: Health Services Research
Other Study IDs: 833396; 4R33AG057380-03 (NIH)
Record Dates: First submitted 2020-03-10; First posted 2020-03-13 (Actual); Last update posted 2021-05-21 (Actual); Status verified 2021-05

CONDITIONS: Cardiovascular Diseases
Keywords: Statin
MeSH Terms: conditions — Cardiovascular Diseases

STUDY DESIGN:
Intervention Model Description: The four-arm factorial trial will randomly assign primary care practices to one of the following arms for the intervention:
  1. Control
  2. Clinician nudge using an active choice prompt in the electronic health record at the time of the patient visit and a monthly peer comparison message on statin prescribing performance relative to peer clinicians at Penn Medicine delivered through the electronic health record
  3. Patient nudge using a text message sent 72 hours prior to their primary care clinician appointment that informs them of their eligibility for a statin, the risks and benefits, and asking them to discuss the role of starting a statin with their clinician
  4. Both clinician nudge and patient nudges
Who Masked: Investigator, Outcomes Assessor
Masking Description: Investigators, statisticians, and analysts will be blinded during the intervention and analysis. Study staff (project director, manager, and research coordinators) will be unblinded throughout the study in order to deliver the appropriate interventions and to manage participant communications. The project manager will be tasked with maintaining codes to associate the blinded assignments to the clinical practices.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Control (No Intervention): Control arm will receive no intervention.
- Clinician nudge (Experimental): The clinician nudge using an active choice intervention in the electronic health record will be delivered to the clinician during the patient's visit. This will be through a Best Practice Advisory that describes the guideline criteria for which the patient is eligible for statin therapy, provides pre-selected options for a statin with alternative options.
  The clinician nudge using monthly peer comparison messages will be sent as an inbox message through the electronic health record. Clinicians will be told what percent of their eligible patients have been prescribed a statin and how that compares to peer clinicians at Penn Medicine.
  Interventions: Behavioral: Clinician Nudge
- Patient nudge (Experimental): The patient nudge will be a text message. Patients with a visit scheduled with their primary care clinician will be identified and sent this text 72 hours before their scheduled visit. The text will remind them of the visit, inform them of their eligibility for a statin, describe the benefits and risks of statin therapy, and ask the patient to discuss statin therapy with their primary care clinician during the visit.
  Interventions: Behavioral: Patient Nudge
- Clinician Nudge and Patient Nudge (Experimental): The clinician nudge and patient nudge will be implemented.
  Interventions: Behavioral: Clinician Nudge; Behavioral: Patient Nudge

INTERVENTIONS:
Behavioral: Clinician Nudge — Active choice intervention in the electronic health record and peer comparison messaging on performance
  Arms: Clinician Nudge and Patient Nudge; Clinician nudge
Behavioral: Patient Nudge — Text message sent to patients to prompt awareness of statin eligibility before an appointment with their primary care physician
  Arms: Clinician Nudge and Patient Nudge; Patient nudge

SUMMARY:
The objective of the study is to evaluate the effect of nudges to clinicians, patients, or both to initiate statin prescriptions for patients that meet national guidelines.

DETAILED DESCRIPTION:
Cardiovascular disease (CVD) is the leading cause of mortality in the United States. Statins have been demonstrated to be an effective tool for reducing the risk of CVD-related events and mortality, but statins are often not prescribed for patients that meet evidence-based guidelines. In this study, the investigators will evaluate nudges to clinicians, patients, or both to initiate statin prescriptions for patients that meet the United States Preventive Task Force guidelines, patients with clinical atherosclerotic cardiovascular disease (ASCVD) condition, and patients with a history of familial hyperlipidemia. In partnership with the health system, this will be conducted as a 4-arm factorial, cluster randomized trial to evaluate the effect of the interventions.

ELIGIBILITY:
Inclusion Criteria:

1. Have new or return visit with a primary care provider at one of the study practices at the University of Pennsylvania Health System
2. Either have an ASCVD condition, history of familial hyperlipidemia, or meet United State Preventive Task Force Guidelines for Statin Therapy which includes age 40-75 years, at least 1 cardiovascular risk factor (e.g. dyslipidemia, diabetes, hypertension, smoking), 10-year ASVCD risk score ≥ 10%

Exclusion Criteria:

1. Already prescribed a statin
2. Allergy to statins
3. Severe renal insufficiency defined as glomerular filtration rate (GFR) less than 30 mL/min or on dialysis
4. Adverse reaction to statins including statin-related a) myopathy; b) Rhabdomyolysis; c) hepatitis
5. Pregnant
6. Currently breastfeeding
7. on hospice or at the end-of-life
8. On a PCSK9 Inhibitor medication

Clinicians (and their respective patients) will be excluded if they have less than 10 patients among their entire panel that are eligible for a statin medication.

Ages: 21 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4131 (Actual)
Dates: Start 2020-10-19 (Actual); Primary Completion 2021-04-18 (Actual); Study Completion 2021-04-18 (Actual)

PRIMARY OUTCOMES:
Statin Prescribing | 6 months
  Change in percent of patients prescribed a statin medication.

CONTACTS AND LOCATIONS:
Overall Officials: Mitesh Patel, MD, MBA, MS, Principal Investigator — University of Pennsylvania
Locations (1):
- University of Pennsylvania, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: Yes
The study protocol will be submitted as an appendix to the main manuscript for publication in an academic journal. Changes to the electronic health record to implement the intervention will be described in the main study manuscript. If any coding is required, it will be made accessible to other researchers on Dataverse, an open source web application. After publication of the main findings, analytical codes used to process and analyze the data will be made available to other researchers on Dataverse, an open source web application.
Supporting Information: Study Protocol, SAP, Analytic Code
Time Frame: Data and datasets will be kept and available to share for at least three years following completion of the project, in accordance with NIH regulations.
Access Criteria: Because electronic health record data contains sensitive patient information, it will be made available to external investigators and the public on a case-by-case basis, to be approved by Dr. Patel, in accordance with institutional, HIPAA, state and federal regulations. A data-sharing agreement may be instituted, depending upon the data to be shared. All data that is shared will be de-identified to protect participant privacy and confidentiality

REFERENCES:
- [Derived] Adusumalli S, Kanter GP, Small DS, Asch DA, Volpp KG, Park SH, Gitelman Y, Do D, Leri D, Rhodes C, VanZandbergen C, Howell JT, Epps M, Cavella AM, Wenger M, Harrington TO, Clark K, Westover JE, Snider CK, Patel MS. Effect of Nudges to Clinicians, Patients, or Both to Increase Statin Prescribing: A Cluster Randomized Clinical Trial. JAMA Cardiol. 2023 Jan 1;8(1):23-30. doi: 10.1001/jamacardio.2022.4373. PMID 36449275